CLINICAL TRIAL: NCT01916668
Title: A Cross-sectional Study on Intradialytic Hypertension at Four Haemodialysis Units in the Western Cape, South Africa
Brief Title: A Cross-sectional Study on Intradialytic Hypertension at Four Haemodialysis Units in the Western Cape
Status: Completed | Type: Observational
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Mogamat-Yazied Chothia, Consultant Nephrologist, University of Stellenbosch
Other Study IDs: S12/10/264
Record Dates: First submitted 2013-02-01; First posted 2013-08-05 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Intradialytic Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational evidence indicates that intradialytic hypertension is associated with high morbidity & mortality. The investigators impression is that this problem may be more prevalent than initially suspected. To the investigators knowledge, there are no studies on intradialytic hypertension in the South African haemodialysis population.

DETAILED DESCRIPTION:
Introduction

Intradialytic hypertension (IDH) is the paradoxical rise in blood pressure (BP) during or immediately after haemodialysis.

Nephrologists have yet to arrive at a standard definition of IDH. Definitions vary widely from systolic blood pressure rises of ≥ 10mmHg, rise in mean arterial pressure (MAP) during dialysis > 15mmHg to hypertension that appears resistant to ultrafiltration during or immediately after dialysis.1 Depending on the definition used, the prevalence of IDH varies between 5-15%.

This phenomenon may appear trivial to the inexperienced doctor. However, IDH increases the risk of hospitalization and death as reported in the Crit-Line Intradialytic Monitoring Benefit Study (CLIMB) and United States Renal Data System (USRDS) haemodialysis study.

The pathogenesis of IDH is unclear. A number of factors have been implicated and probably work synergistically to promote the rise in BP. These include: subclinical volume overload, activation of the sympathetic and renin-angiotensin-aldosterone systems, endothelial dysfunction, sodium gain during dialysis, use of erythropoietin stimulating agents (ESAs) and removal of anti-hypertensive agents during dialysis.

The management of IDH relies heavily on control of sodium and fluid dynamics. There are no randomized controlled studies to guide management.

Objectives

Primary: Determine the prevalence of IDH at four haemodialysis units in the Western Cape

Secondary: To examine the association between IDH and the following potential risk factors:

Intradialytic weight gain, the presence and/or degree of fluid overload as assessed by bioimpedance monitoring, quantity and timing of anti-hypertensive drugs, ESA dose and route of administration, time-averaged sodium concentration, dialysate calcium concentrations and haemodialysis modality.

Methods

Study Design

A multicentre, cross-sectional study on chronic haemodialysis patients at four adult dialysis units in the Western Cape will be conducted.IDH will be defined as a rise of ≥10mmHg in systolic blood pressure between pre- and post-dialysis in at least 4 out of six dialysis sessions. Patients screened as eligible for inclusion in the study will be identified from haemodialysis charts by the primary investigator (PI). They will then be approached by the PI, who will try to obtain informed consent. Once informed consent has been obtained and no exclusion criteria are present, the patient will be enrolled. A study ID number will be allocated.

Using a standard operating protocol (SOP), weight, BP, pulse rate, bioimpedance, ultrafiltration rates and volumes will be determined before, hourly during dialysis and 30 minutes after completion of dialysis. Timing and use of antihypertensive drugs, ESA use, dialysis modality, intradialytic calcium and time averaged sodium levels will be determined. All data extracted will be captured onto a standardised data sheet.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age > 18 years
* Ability to give informed consent

Exclusion Criteria:

* Inability to take blood pressure by routine methods in the upper limbs
* Inability to give informed consent
* Contraindications to bioimpedance monitoring (pre-existing implanted cardiac devices such as pacemakers, cardioverter defibrillators; amputees)
* Intercurrent acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic haemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of intradialytic hypertension at four haemodialysis units in the Western Cape | Up to 1 year

SECONDARY OUTCOMES:
Participants pre- and post hemodialysis bioimpedance measurements | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mogamat-Yazied Dr Chothia, FCP(SA), Principal Investigator — University of Stellenbosch
Locations (1):
- Tygerberg Academic Hospital, Cape Town, Western Cape, South Africa